CLINICAL TRIAL: NCT00523484
Title: An Observational Study to Assess Correlation Between Prostate Specific Antigen & Beck Anxiety Index in Prostate Cancer Patients Under Hormonal Therapy
Brief Title: Casodex/Zoladex Hormonal therApy Study for assessMent of Correlation Between PSA & BAI in prOstate Cancer patieNts
Acronym: CHAMPION
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC CD, AstraZeneca
Other Study IDs: NIS-OKR-CAS-2007/1
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Prostate Cancer
Keywords: Beck Anxiety Inventory; Prostate Cancer; Prostate Specific Antigen; Naturalistic; Observational
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an observational study to see whether anxiety level can be correlated with PSA level under the current practice in the patients of prostate cancer taking hormonal therapy. For assessment of anxiety level BAI(Beck Anxiety Inventory) will be used. The target population for this study is the patients of prostate cancer diagnosed previously and who are taking hormonal therapy with regular follow-up and PSA test. The follow-up duration will be total 6 months with interim visit at 3 month and final visit at 6 month.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Patients who take PSA test regularly
3. Observation suitable patients for PSA change according to hormonal treatment at least for 6months
4. Locally advanced or advanced prostate cancer patients who is suitable for hormonal therapy
5. Prostate Cancer Patients who has been taking one treatment among 3 hormonal therapies in below:

   * Bicalutamide Monotherapy : Bicalutamide 150mg/day
   * Goserelin 3.6mg/10.8mg
   * MAB(Maximal Androgen Blockade) :Bicalutamide 50mg + Goserelin 3.6/10.8mg

Exclusion Criteria:

1. Prohibition use under permitted indication
2. Previous inclusion in the present study
3. Participation in a clinical study during the last 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced prostate cancer patients who were being treated by hormonal agents
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miyoung Kim, Study Director — AstraZeneca Korea
Locations (3):
- South Korea (3):
  - Research Site, Kyunggi, Anyang-si Dongan-gu
  - Research Site, Seoul, Jongro-gu
  - Research Site, Seoul, Songpa-gu